CLINICAL TRIAL: NCT06939634
Title: Evaluation of Usability and Safety of the System Atalante in Patients With High Paraplegia and Tetraplegia
Acronym: QUATRO
Status: Completed | Type: Observational
Sponsor: Wandercraft (Industry)
Responsible Party: Sponsor
Other Study IDs: CIP009
Record Dates: First submitted 2025-03-04; First posted 2025-04-23 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-03

CONDITIONS: Spinal Cord Injury; Tetraplegia/Tetraparesis; Paraplegia, Complete; Paraplegia, Incomplete; Guillain Barré Syndrome
Keywords: Hands-free Exoskeleton; Atalante X; Atalante; Rehabilitation; Safety
MeSH Terms: conditions — Spinal Cord Injuries; Quadriplegia; Paraplegia; Guillain-Barre Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Hands-free exoskeleton: Patient with high paraplegia or tetraplegia who have undergone at least one session with the exoskeleton.
  Interventions: Device: Hands-free exoskeleton

INTERVENTIONS:
Device: Hands-free exoskeleton — Having undergone at least on session with Atalante exoskeleton. Clinical, safety and session data are collected retrospectively.

SUMMARY:
The objective of this clinical trial is to determine whether the Atalante X exoskeleton can be safely utilized by patients with tetraplegia and high paraplegia (at or above T4).

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old,
* Tetraplegia or high paraplegia (at or above T4) regardless of the cause,
* Non-opposition to the participation to the study,
* Having undergone a minimum of 1 session with the Atalante device from February 2019, to now.

Exclusion Criteria:

* Neurological Level of Injury below T4 as determined by the International Standards for Neurological Classification of SCI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population includes people with high paraplegia and tetraplegia.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Safety through the collection of the reported adverse device effects | Baseline, up to 101 weeks.
  Measured through all reported adverse device effects (ADEs). ADEs are categorized into the following categories: musculoskeletal, cutaneous (skin abrasion), cardiovascular (orthostatic hypotension), pain, falls, and fractures and are further characterized as minor or serious based on the nature and the severity of the adverse event (AE).

SECONDARY OUTCOMES:
Spasticity assessment | Baseline, post-intervention (up to 101 weeks)
  This may involve the use of the Modified Ashworth Scale or a general description of spasticity recorded in the medical file.
Walking ability | Baseline, post-intervention (up to 101 weeks)
  This may involve Walking Index for Spinal Cord Injury, version II (WISCI II) assessing the amount of physical assistance needed, as well as devices required, for walking following paralysis that results from SCI. It ranges from 0 (unable to stand and/or participate in assisted walking) to 20 (ambulates with no devices, no braces and no physical assistance, 10 meters).
Walking speed | Baseline, post-intervention (up to 101 weeks)
  This may involve 10 meters walk test (10MWT) measuring gait speed during a 10-meter walk during comfortable and rapid pace.
Mobility, balance, walking ability, and fall | Baseline, post-intervention (up to 101 weeks)
  This may involve Time Up and Go (TUG), a timed task where the patient is asked to stand up from the chair, walk 3 meters, turn around, walk and sit again.
Endurance | Baseline, post-intervention (up to 101 weeks)
  This may involve 6-minutes' walk test (6MWT) and 2-minutes' walk test (2MWT) measuring the walked distance during a 6- or 2-minutes' walk.
Balance | Baseline, post-intervention (up to 101 weeks)
  This may involve Berg Balance Scale (BBS) including items include static and dynamic activities of varying difficulty.
Independance | Baseline, post-intervention (up to 101 weeks)
  This may involve Spinal Cord Independence Measure (SCIM III) including items assessing self-care, respiration and sphincter management.
Usability assessment | Post-intervention (up to 101 weeks)
  The assessment of the usability will be asked to the operators in charge of the rehabilitation of the patients included in this study. It includes a usability questionnaire and session data collection.

OTHER OUTCOMES:
Descriptive data: Age | Baseline, up to 101 weeks.
  To characterize the population, for each patient, the age will be collected when available (years).
Descriptive data: Gender | Baseline, up to 101 weeks.
  To characterize the population, for each patient, the gender will be collected when available (male, female).
Descriptive data: Cause and time since injury or pathology | Baseline, up to 101 weeks.
  To characterize the population, for each patient, the cause of injury or pathology, the time since injury or diagnosis (years) will be collected when available.
Descriptive data: Urinary status | Baseline, up to 101 weeks.
  To characterize the population, for each patient, the urinary status will be collected when available:
  * Intermittent catherization
  * Indwelling catherization
  * External collection device
  * Other
Descriptive data: Bowel status | Baseline, up to 101 weeks.
  To characterize the population, for each patient, the bowel status will be collected when available:
  * Digital stimulation
  * Manual evacuation
  * Colostomy
  * Other
Descriptive data: Severity of the lesion using the International Standards for Neurological Classification of SCI | Baseline, up to 101 weeks.
  To characterize the population, for each patient, the following descriptive data will be collected when available:
  * ASIA impairement scale: A (complete), B (sensory incomplete), C and D (motor incomplete), E (normal).
  * Neurological Level of Injury
Descriptive data: Cardiorespiratory parameters | Baseline, up to 101 weeks.
  To characterize the population, for each patient, cardiorespiratory parameters including Heart Rate (HR) in Beats per minute and Blood Pressure (BP) in mmHg will be collected when available.
Descriptive data: Pain | Baseline, up to 101 weeks.
  To characterize the population, for each patient, intensity of the pain using the subjective Numeric Pain Rating Scale (NPRS) will be collected when available: from 0 (no pain) to 10 (worst possible pain).
Descriptive data: Bone health | Baseline, up to 101 weeks.
  To characterize the study population, bone health data will be collected for each patient, when available, including:
  * T-score values ranging from 0 (normal) to below -2.5 (indicative of osteoporosis)
  * Bone Mineral Density (BMD) measurements expressed in g/cm²
Reasons for discontinuing sessions | Post-intervention (up to 101 weeks)
  The reason(s) for discontinuing sessions may include hospital discharge, patient's decision, pain or discomfort, achievement of goals set by the therapeutic team, etc.

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Fondation Hopale, Berck, France
  - CMPR de Pionsat, Pionsat, France
  - Hôpital La Musse, Saint-Sébastien-de-Morsent, France

IPD SHARING:
Plan to Share IPD: No